CLINICAL TRIAL: NCT05512988
Title: A Randomized, Double-blind, Controlled Clinical Study of Human Umbilical Cord Mesenchymal Stem Cell(UC-MSC)Delayed Renal Chronic Kidney Disease(CKD3、4 )
Brief Title: Human Umbilical Cord Mesenchymal Stem Cell(UC-MSC)Delayed Renal Chronic Kidney Disease(CKD3、4 )
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Zhongyuan Xiehe Biological Cell Storage Service (Tianjin) Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Gang Xu, Principle Investigator, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TongjiHospitalxugangtjh
Record Dates: First submitted 2022-08-18; First posted 2022-08-23 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Diseases; human umbilical cord Mesenchymal stem cell; CKD3/CKD4
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): MSCs Participants will receive HUC-MSCs
  Interventions: Biological: UC-MSC
- Comparator (Placebo Comparator): Comparator participants will receive saline solution
  Interventions: Biological: Saline solution

INTERVENTIONS:
Biological: UC-MSC — Usage: The stem cell preparation in this study is used intravenously in the elbow.
  Dose: The dose of stem cell injection in this clinical study is set at 1×10^6/Kg/time per injection, and the injection frequency is 2 weeks/time.
  Duration: 2 injections per trial group for the entire duration of the course, with a total dose of 2×10^6/Kg/person.
  Arms: Experimental
Biological: Saline solution — Usage: The saline solution in this study is used intravenously in the elbow.
  Dose: The dose of saline solution in this clinical study is set at 250ml/time per injection, and the injection frequency is 2 weeks/time.
  Duration: 2 injections per person for the entire duration of the course
  Arms: Comparator

SUMMARY:
The chronic kidney disease is caused by renal structural and functional impairment for more than 3 months due to various causes, including normal and abnormal glomerular filtration rate (GFR), abnormal blood, urine, and imaging findings, or an unexplained decline in GFR (<60 ml/min). Recent years, the incidence of chronic kidney disease has increased year by year worldwide, the incidence of CKD is 8% to 16% in the world's total population. chronic kidney disease has become an important public health problem in China and even the world.

Summarizing the basic and clinical studies at home and abroad, inflammatory factors such as inflammatory chemokines, cytokines, and reactive oxygen species interact with fibrosis factors such as mesangial cells, fibroblasts, and fibroblast activation, which are the root causes of the progression of CKD and the formation of tubular interstitial fibrosis and glomerular sclerosis and developing into end-stage renal disease.

Current treatments for chronic kidney disease are very limited, and to be precise, there is currently no cure for chronic kidney disease, nor is there a proven way to improve the kidneys survive after acute kidney injury (AKI). The progression of the disease itself can only be delayed as much as possible by changing the diet, controlling related complications with oral medications (such as hypertension, hyperlipidemia, nephropathy, etc.), and actively controlling blood glucose and glycosylated hemoglobin levels in patients with diabetes. For patients with stage CKD5 and more severe, renal replacement therapy is recommended, including hemodialysis and peritoneal dialysis, but there are many complications in both dialysis methods, such as narrowing of the internal fistula, occlusion, catheter infection, peritonitis, etc. Kidney transplantation may be considered when economic conditions permit and there is a matching kidney source, but kidney transplant surgery is riskier. The above treatment methods have brought a heavy burden to patients and social medicine. In order to seek innovative and effective strategies to cultivate the limited regenerative capacity of the kidneys and reverse renal fibrosis, the mesenchymal stem cells (MSCs) with tissue regenerative potential and immunomodulatory functions have brought new ideas and hopes for the prevention and treatment of chronic kidney disease.

DETAILED DESCRIPTION:
The chronic kidney disease is caused by renal structural and functional impairment for more than 3 months due to various causes, including normal and abnormal glomerular filtration rate (GFR), abnormal blood, urine, and imaging findings, or an unexplained decline in GFR (<60 ml/min). Recent years, the incidence of chronic kidney disease has increased year by year worldwide, the incidence of CKD is 8% to 16% in the world's total population. The incidence of CKD and the primary causative factors vary from country to country and region, and the idemiological survey led by Peking University Hospital shows that the prevalence of CKD in China is 10.8% , the primary causative factor is glomerulonephritis, but as the incidence of hypertension and diabetes rises year by year, and the world will have more than 10 million people a year have acute kidney injury, the proportion of chronic kidney disease in the long-term course of the above population will be much higher than the normal population, chronic kidney disease has become an important public health problem in China and even the world.

Summarizing the basic and clinical studies at home and abroad, inflammatory factors such as inflammatory chemokines, cytokines, and reactive oxygen species interact with fibrosis factors such as mesangial cells, fibroblasts, and fibroblast activation, which are the root causes of the progression of CKD and the formation of tubular interstitial fibrosis and glomerular sclerosis and developing into end-stage renal disease.

Current treatments for chronic kidney disease are very limited, and to be precise, there is currently no cure for chronic kidney disease, nor is there a proven way to improve the kidneys survive after acute kidney injury (AKI). The progression of the disease itself can only be delayed as much as possible by changing the diet, controlling related complications with oral medications (such as hypertension, hyperlipidemia, nephropathy, etc.), and actively controlling blood glucose and glycosylated hemoglobin levels in patients with diabetes. For patients with stage CKD5 and more severe, renal replacement therapy is recommended, including hemodialysis and peritoneal dialysis, but there are many complications in both dialysis methods, such as narrowing of the internal fistula, occlusion, catheter infection, peritonitis, etc. The presence of the above complications will reduce the service life of the patient's dialysis pathway while also causing blows to other organ systems. Kidney transplantation may be considered when economic conditions permit and there is a matching kidney source, but kidney transplant surgery is riskier, and the average survival of transplanted kidneys is currently 12 years calculated by the American National Kidney Foundation, during this period, patients need to take anti-rejection drugs uninterruptedly, and these drugs (such as tacrolimus, cyclosporine, etc.) can also greatly damage the kidney organs and function. The above treatment methods have brought a heavy burden to patients and social medicine. In order to seek innovative and effective strategies to cultivate the limited regenerative capacity of the kidneys and reverse renal fibrosis, the mesenchymal stem cells (MSCs) with tissue regenerative potential and immunomodulatory functions have brought new ideas and hopes for the prevention and treatment of chronic kidney disease.

Progression in chronic kidney disease includes tubular interstitial fibrosis and glomerulosclerosis:

1) Tubular interstitial fibrosis is mainly characterized by tubular hypermetabolism, tubular epithelial-interstitial transition, and hypoxic damage to the renal interstitium, which eventually leads to infiltration of inflammatory cells, abnormal increase in extracellular matrix components in renal tissue, and disappearance of parenchymal cells. 2)Glomerulosclerosis is the outcome of excessive response of glomerular constituent related cells to injury, including structural changes, cells' gradual atrophy, shedding, apoptosis of cells, loss of anticoagulant properties, and increased expression of pro-inflammatory factors and pro-fibrosis factors; Proliferation of mesangial cells, mesangial differentiation into myofibroblasts, causing collagen III to be deposited in the renal units, leading to irreversible hardening of the glomeruli; The number of pinus process cells decreases, the skeleton retracts or flattens, and inflammatory cell aggregation of chemokines is released, while synthetic cytokines and growth factors further aggravate globules capillary sclerosis.

Both pathophysiological abnormalities are characterized by parenchymal cell loss and activation of the inflammatory immune response. However, due to the weak regenerative capacity of renal tubular epithelial cells and endothelial cells, foot process cells even lack regenerative ability, these renal parenchymal cells are difficult to repair themselves once damaged, and the kidney lacks stem/progenitor cells, which cannot achieve stem/progenitor cell differentiation and regeneration. Therefore, after severe kidney damage, the existing treatment methods cannot promote the complete repair of the kidneys, often resulting in the delay of kidney disease, which is also the main reason why chronic kidney disease has become the highest incidence of chronic disease in humans.

MSCs are only briefly present in the renal vascular system, and Togel F, Hu Z et al. found that their presence was not detected within the renal parenchyma after 3 days of MSC infusion, and in general, stem cells were only briefly present in the blood vessels of the kidneys and could not colonize for long periods of time7. Studies such as Camila Eleuterio Rodrigues found that gene expression in the kidneys of MSC-treated rats showed a decrease in pro-inflammatory cytokines and an increase in several growth factors with pro-mitosis, pro-survival, and anti-apoptosis effects8. There is a large body of research evidence that MSCs modulate the immune response primarily through paracrine/endocrine nutritional growth factors and ultimately promote renal repair.1)Stem cells secrete immunomodulatory correlates;2) Stem cell secretion promotes renal vascular formation and tubular cell regeneration related factors;3)MSC may also reduce renal fibrosis and structural remodeling through immunomodulation;4)Stem cell secretion improves matrix metabolism-related factors.

mesenchymal stem cell therapy has a good safety record, there is no obvious toxic side effects for patients, a small number of patients have injection of local discomfort, transient low-grade fever, etc., generally do not need special treatment, patients will recover naturally, long-term observation has not found that patients have increased microbial infections and the carcinogenicity of Mesenchymal stem cell.

Characteristics and advantages of umbilical cord mesenchymal stem cells, MSCs isolated from umbilical cord tissue, not only maintain the biological characteristics of MSCs, but also have the following advantages compared to other tissue-derived mesenchymal stem cells: 1) Convenient materials, which is waste utilization. 2) The process is less invasive to the donor than the extraction of bone marrow MSCs. 3) The isolated cell content and proliferation ability are better than bone marrow MSCs, and the immunogenicity is lower than that of bone marrow MSCs, which is not easy to trigger the immune response or cause graft-versus-host disease. 4) The differentiation potential is stronger, and differentiation can be carried out in multiple directions. 5) Stronger ability to secrete cytokines and may have a stronger paracrine (exosome) repair effect. 6) Compared with bone marrow MSCs, the results of gene lineage comparison show that umbilical cord mesenchymal stem cells can express more genes and proteins related to matrix remodeling and angiogenesis, which is more suitable in the field of nephropathy treatment.

Therefore, in the field of nephropathy treatment, umbilical cord MSC has greater potential for application.

This study was a prospective, single center, randomized controlled and double-blind study, total duration 36 months, of which each patient study cycle is 13 months, and long-term safety follow-up is 12 months after the end of the study. It is grouped by the random number table method, divided into the experimental group and the control group according to the ratio of 1:1, 22 people were required in the experimental group and 22 people in the control group, for a total of 44 people. Experimental group will receive UC-MSC, while the control group will receive saline solution. The expected effect is UC-MSC can delay the progression of renal function in patients with brady nephropathy,reduced or alleviated chronic kidney disease-related complications (e.g., anemia, hypertension).

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of chronic kidney disease (CKD) and stage 3 and stage 4 (GFR 15-60 ml/min) of CKD (American Kidney Disease Foundation stage)
* Agree to sign the informed consent form at the same time by means of participation of the pilot group
* Age between 18-65 years old

Exclusion Criteria:

* Patients who are taking immunosuppressants or have been taking them within a month
* Patients with a 30% increase in creatinine in the past 3 months and who are about to undergo dialysis
* Suffering from severe heart, respiratory insufficiency, viral hepatitis, and sexually transmitted diseases
* Hypersensitivity to stem cells themselves or stem cell-related media
* Patients with recent bacterial, viral, or fungal infections
* Have a history of tumors or are currently suffering from tumor conditions
* Pregnant or breastfeeding
* Have participated in drug-related clinical trials in the past two months
* Any form of substance abuse, mental illness, and other conditions that researchers believe may affect the effectiveness of the test or the patient's physical health

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-04-13 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change of GFR | baseline, 6-month after 2nd treatment, 12-month after 2nd treatment
  GFR decrease at 2.5ml/min/year or more from baseline
Incidence of Treatment-Serious Adverse Events as assessed by SPSS 23.0 and Graphpad prism 6 | Through study completion, an average of 13 months
  To observe the incidence of serious adverse events，such as fatal cardiovascular and cerebrovascular disease, tumor, organ failure, severe infection.
Number of participants with treatment-related adverse events as assessed by SPSS 23.0 and Graphpad prism 6 | Through study completion, an average of 13 months
  Collecting and comparing the number and severity of participants with skin reactions, fever, infection, allergic reactions, etc. in the two groups.

SECONDARY OUTCOMES:
IgA | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  Change of humoral immunity after stem cell treatment
IgG | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  Change of humoral immunity after stem cell treatment
IgM | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  Change of humoral immunity after stem cell treatment
C3 | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  Change of humoral immunity after stem cell treatment
C4 | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  Change of humoral immunity after stem cell treatment
CRP | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  Changes in inflammatory and immunological serologic indicators after stem cell treatment
IL-6 | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  Changes in inflammatory and immunological serologic indicators after stem cell treatment
Peripheral hemolymocyte subsets | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  Changes in inflammatory and immunological serologic indicators after stem cell treatment
Urine protein | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  To observe the change of urine test after stem cell treatment
Urine RBC | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  To observe the change of urine test after stem cell treatment
24-hour urine protein | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  To observe the change of urine test after stem cell treatment
Urine albumin/creatinine | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  To observe the change of urine test after stem cell treatment
Electrolytes | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  The change of electrolytes was detected after treatment
Hemoglobin | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  The change of hemoglobin was detected after treatment
Albumin | 2 weeks after the first treatment, 1 month, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  The change of albumin was detected after treatment
Heart ultrasound | Baseline, 3 months, 6 months and 9 months, 12 months,18 months, 24 months after the second treatment
  To assess the incidence of complications in other organ systems, such as cardiovascular, skeletal, and hematopoietic systems
Carotid ultrasound | Baseline, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  To assess the incidence of complications in other organ systems, such as cardiovascular, skeletal, and hematopoietic systems
NT-proBNP | Baseline, 2nd treatment, 1 months, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  To assess the incidence of complications in other organ systems, such as cardiovascular, skeletal, and hematopoietic systems
iPTH+1,25-VitD3 | Baseline, 2nd treatment, 1 months, 3 months, 6 months and 9 months, 12 months, 18 months, 24 months after the second treatment
  To assess the incidence of complications in other organ systems, such as cardiovascular, skeletal, and hematopoietic systems

CONTACTS AND LOCATIONS:
Overall Officials: GANG XU, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
After approval from the steering committee and the Human Genetic Resources Administration of China, this trial data can be shared with qualifying researchers who submit a proposal with a valuable research question. A contract should be signed.